CLINICAL TRIAL: NCT05399576
Title: The Preventive Effect of Combined Intracoronary of Nicorandil and Verapamil on Myocardial Injury in Preioperative Period of PCI
Brief Title: Intracoronary of Nicorandil and Verapamil to Reduce the Occurrence of Periprocedural Myocardial Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-KL-085-03
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: periprocedural myocardial injury; coronary microvascular disturbances; percutaneous coronary intervention; nicorandil; verapamil
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nicorandil; Verapamil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicorandil and verapamil (Experimental): intracoronary of 2mg Nicorandil and 500ug verapamil
  Interventions: Drug: Nicorandil
- saline (Placebo Comparator): intracoronary of 4ml saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nicorandil — Prophylactically combined intracoronary of Nicorandil and verapamil
  Other Names: verapamil
  Arms: Nicorandil and verapamil
Drug: Saline — intracoronary of 4ml saline
  Arms: saline

SUMMARY:
Percutaneous coronary intervention (PCI) remains the major revascularization strategy for patients with obstructive coronary artery disease (CAD).However,in a substantial number of PCI cases for acute coronary syndrome (ACS) and chronic coronary syndrome (CCS),periprocedural myocardial injury or myocardial infarction (MI) occurs,both these PCI-related complications may be associated with an increased risk of future major adverse cardiovascular events (such as death, re-infarction, and revascularization).The incidence of periprocedural myocardial injury varies according to the different definition and cardiac biomarker .For 4th UDMI criteria with hs-cTn, 78% to 85% patients who undergoing elective PCI may suffer from periprocedural myocardial injury.

Experimental and clinical evidence highlight the abnormalities of the coronary microcirculation is one of the causes of myocardial ischemia.Coronary microvascular disturbances (CMD) have been associated with early stages of atherosclerosis even prior to any angiographic evidence of epicardial coronary stenosis, as well as to other cardiac pathologies such as myocardial hypertrophy and heart failure.

In this study, we try to conduct a double blinded, randomized, placebo-controlled trial，the aim of our trial is: (1) to observe whether the prophylactically intracoronary administration of nicorandil and verapamil could reduce the occurrence of periprocedural myocardial injury and infarction in CAD patients undergoing elective PCI.;(2) to observe whether the prophylactically intracoronary administration of nicorandil and verapamil has protective effect on coronary microcirculation after elective PCI.

DETAILED DESCRIPTION:
Simple randomization in a 1:1 ratio will be made in blocks of variable size according to a random numbers generated by Excel 2019 to divide the patients to treatment group (Nicorandil and verapamil) and control group (Saline). The primary end points are the incidence of periprocedural myocardial injury and 4a MI and the level of the IMR,secondary end points include levels of hs-cTnI, CK-MB ,NT-proBNP and hs-CRP before, and 24 hours following PCI, and major adverse cardiovascular events at day 30. SPSS 26.0 will be used, and P-value < .05 will be considered statistically signifificant.

ELIGIBILITY:
Inclusion Criteria:

* 1.diagnosis of CHD with FFR<0.8;2.elective PCI;

Exclusion Criteria:

* Patients with AMI, lesion at the opening of the main coronary artery，kidney dysfunction, Liver dysfunction，blood coagulation disorder ,NYHA III-IV,Degree II-III atrioventricular block,and restenosis after PCI，CABG will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-05-17 (Estimated); Study Completion 2023-09-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of periprocedural myocardial injury and infarction after PCI | Within 24 hours after surgery
  2.periprocedural myocardial injury was defined as hypersensitive troponin exceeding the upper limit of normal after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- yuangang Qiu, Hangzhou, Zhejiang, China